CLINICAL TRIAL: NCT06775639
Title: Should we Avoid Performing Invasive Coronary Angiography Before Cardiac Surgery in ACHD (Adult Congenital Heart Disease) Patients? The SPARE Observational Study
Brief Title: Should we Avoid Performing Invasive Coronary Angiography Before Cardiac Surgery in ACHD Patients?
Acronym: SPARE
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: SPARE
Record Dates: First submitted 2024-11-28; First posted 2025-01-15 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2024-10

CONDITIONS: Adult Congenital Heart Disease
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to compare two pre-operative methods, that is the Invasive Coronary Angiography (ICA), an actual standard diagnostic method, with the Coronary Computer Tomography (CCT) to undestand if the only CCT is sufficent to confirm the presence of a significative coronary disease and so to identify possible lesions in the coronary ematic circle, for example: stenosis and narrowing of coronary vessels. This observational study included people who have a congenital heart desease with indication of cardiac surgery and, why this disease, who had already performed these two diagnostic methods and/or who will perform them. The main question it aims to answer is: Should we avoid performing invasive coronary angiography (ICA) before cardiac surgery in people who have congenital heart desease (ACHD patients)?

DETAILED DESCRIPTION:
The primary aim is to verify the diagnostic reliability of coronary CCT to confirm or exclude the presence of significant coronary artery disease in ACHD patients who are candidates for cardiac surgery compared to ICA, the current gold standard.

the Secondary objectives is to measure the occurrence of side effects and/or complications secondary to ICA and CCT procedures. To measure the frequency with which each of the two methods is able to identify the presence of coronary anomaly and the correct anatomical relationships between the anomalous coronary artery and the adjacent structures. To compare the waiting times of coronary CCT and coronarography, in order to assess their actual availability in daily clinical practice.

The primary outcomes of the study are:

* non-significant lesions of the coronary tree (stenosis < 50%)
* significant lesions (stenosis ≥ 50%)
* limited to CCT investigation: coronary tree partially or completely unassessable due to artefacts or extensive calcifications preventing proper assessment.

ELIGIBILITY:
Inclusion Criteria:

* Adult congenital heart disease patient who is a candidate for cardiac surgery for correction of defect valve, or who performed the surgery after 01.01.2010
* Clinical indication for preoperative ICA and CCT performed less than 12 months apart within 12 months of planned cardiac surgery
* Age ≥ 18 years
* Obtaining written informed consent

Exclusion Criteria:

* Inability to perform ICA for any reason (e.g., poor vascular access or anatomical difficulty in reaching the coronary arteries)
* Patient with severe renal failure on dialysis therapy
* Patient with previous cerebri stroke

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study will include ACHD patients referred to the Pediatric Cardiology and Cardiac Surgery of the Cardiology Operating Unit of the IRCCS AOU of Bologna, candidates for surgery cardiac surgery with clinical indication to undergo preoperative ICA and CCT. The SPARE study will include only patients with independent clinical indication to CCT.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-01-08 (Estimated); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Non-significant and significant coronary lesions | Immediately after the procedure
  Coronary lesions will be defined as nonsignificant when they result in a narrowing of the lumen of the coronary artery less than 50%. Lesions will be considered significant when they will result in a narrowing of the lumen of the coronary artery equal to or greater than 50%.
Coronary tree partially or completely unassessable for artifacts or extensive calcifications that prevent proper evaluation | immediately after the procedure
  A portion or the entire coronary tree will be defined as unassessable when it is not it is possible to determine the percentage of stenosis in a coronary segment or in the entire coronary artery.

SECONDARY OUTCOMES:
Side effects/complications from administration of iodinated contrast medium for the performance of Coronary Computer Tomography (CCT) or Invasive CoronaryAngiography (ICA) | Within 48 hours of the investigation.
  Creatininemia elevation of 0.3 mg/dl within 48 hours after surgery, or more than 150% of the initial value or a reduction of diuresis below 0.5 ml/Kg for more than 6 hours. Incidence of cardiac death, heart attack myocardial infarction, stroke, vascular complications and nonvascular at the site of access ie. finding of vascular aneurysm or pseudoaneurysm or obstruction of the artery used for ICA, major bleeding defined as of grade 3 or higher according to the BARC classification.
Identification of abnormal origin from the aortic wall of any of the three major coronary arteries (right coronary artery, anterior interventricular branch, branch circumflex); identification of a different than normal course of any of the three main | At the end of CCT and ICA
  Abnormal origin: finding of abnormal position compared to the normal anatomical position of the ostium of at least one of the coronary arteries (right coronary artery, common trunk or anterior interventricular branch and branch circumflex). Abnormal course: different than normal course of one of the three major arteries coronary arteries. Dangerous course: course through the large vessels (aorta and pulmonary artery or other paracardiac) of one of the three major coronary arteries.
Waiting time for the execution of the of the investigation defined as: time that elapses between the decision to perform CCT and the preoperative ICA | during the procedure
  Interval of time between the decision of the execution of the investigation and the date on which the investigation is conducted

CONTACTS AND LOCATIONS:
Overall Officials: Gabriele Egidy Assenza, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Italy